CLINICAL TRIAL: NCT05978128
Title: Utilizing Spheres of Influence to Increase Cancer Screening: Empowering Community Health Advocates
Brief Title: Utilizing Advocates and Supporters to Increase Lung Cancer Screening Rates in Eligible Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-000947; NCI-2023-04133 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma; Lung Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Health Promotion; Educational Status; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (electronic patient portal, patient navigation) (Experimental): Participants access an electronic patient portal with educational materials at baseline, 1- and 2-year follow-ups, and also interact with a patient navigator on study. Patients also receive materials to share with their friends/family on benefits of breast and lung cancer screening on study.
  Interventions: Behavioral: Health Education; Other: Health Promotion and Education; Behavioral: Patient Navigation; Other: Survey Administration

INTERVENTIONS:
Behavioral: Health Education — Access electronic patient portal with educational material
Other: Health Promotion and Education — Receive materials on breast/lung cancer screening
Behavioral: Patient Navigation — Interact with a patient navigator
  Other Names: Patient Navigator Program
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial assesses the use of advocates and supporters of breast and lung cancer screening to increase lung cancer screening rates amongst eligible participants. Imaging-based cancer screening is utilized with variable frequency. Breast cancer screening with mammography has been widely accepted and is commonly used among eligible women. Lung screening with computed tomography scans is poorly used, despite the potential to decrease deaths from lung cancer. There are many reasons lung screening isn't being used when compared to breast screening, such as smoking stigma and fear, along with a lack of awareness of lung screening. By conducting this trial, researchers want to assess the effectiveness of advocates and supporters of breast and lung screening, and to learn about the psychological barriers to cancer screening, identifying those that are unique to lung screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the number of patients undergoing breast screening who are eligible to participate in lung screening.

II. Determine whether patients currently participating in cancer screening (breast OR lung) are successful as "cancer screening advocates." III. Determine whether laypersons who are aware of screening (including those who accompany friends and family members to their screening appointments) are successful as "cancer screening advocates." IV. Identify knowledge base and psychological barriers to screening through surveys of potential screening participants.

OUTLINE:

Participants access an electronic patient portal with educational materials at baseline, 1- and 2-year follow-ups, and also interact with a patient navigator on study. Patients also receive materials to share with their friends/family on benefits of breast and lung cancer screening on study.

After completion of study intervention, participants are followed up yearly for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age:

  * Breast screening > 40
  * Lung screening 50-80
* Male (M) or Female (F)
* Current, former, or never smokers
* Close family or friend with smoking history (in or out of state)

Exclusion Criteria:

* Age:

  * Breast screening < 40
  * Lung screening < 50 or > 80
* Persons who had previously received a diagnosis of lung cancer, had hemoptysis, or had an unexplained weight loss of more than 6.8 kg (15 lb) in the preceding year will also be excluded
* Persons with an active cancer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Increased rates of lung and breast cancer screening adherence | Up to 3 years
  By following up with patients over the defined study period and assessing whether they obtained an incidence screen completed at one-year +/- 3 months from the recommended time. Will also measure the rates of survey completion by consented participants, the number of clicks and time spent reviewing educational materials, and the number of new participants who contacted the program through a referral by another participant.

SECONDARY OUTCOMES:
Success of "sphere of influence" model | Up to 3 years
  Considered successful if increased lung cancer screening referrals are a direct result of women receiving screening mammograms inviting and educating friends and family about lung cancer screening.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Prosper, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States